CLINICAL TRIAL: NCT07155057
Title: A Prospective, Single-Arm Study Evaluating Crosslinked Hyaluronate Canalicular Gel for the Treatment of Dry Eye Disease in Patients Undergoing Refractive Cataract Surgery
Brief Title: Evaluating Crosslinked Hyaluronate Canalicular Gel for the Treatment of DED in Patients Undergoing Cataract Surgery
Acronym: LaReCa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Lacrifill IIT
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Study Participants (Other): Patients will receive bilateral lacrimal occlusion of crosslinked hyaluronate canalicular gel pre-operatively
  Interventions: Device: Cross-Linked Hyaluronate Gel Prefilled Syringe 30 MG/3ML

INTERVENTIONS:
Device: Cross-Linked Hyaluronate Gel Prefilled Syringe 30 MG/3ML — Prospective, single-site, single-arm study enrolling 60 patients who have elected advanced IOL implantation at the time of cataract surgery and have a diagnosis of dry eye disease. The study will consist of 5 study visits, over a 3-5 month time period. Patients will receive bilateral lacrimal occlusion of crosslinked hyaluronate canalicular gel pre-operatively

SUMMARY:
To review how patients report using a hyaluronate crosslinked canalicular gel placed before cataract surgery

DETAILED DESCRIPTION:
Prospective, single-site, single-arm study enrolling 60 patients who have elected advanced IOL implantation at the time of cataract surgery and have a diagnosis of dry eye disease. The study will consist of 5 study visits, over a 3-5 month time period. Patients will receive bilateral lacrimal occlusion of crosslinked hyaluronate canalicular gel pre-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to understand and sign the informed consent form (ICF)
* Men or non-pregnant women age 22 or older
* Clear intraocular media other than cataract
* Diagnosis of dry eye disease (OSDI score ≥ 13)
* Non-invasive Tear break up time ≤ 10 seconds in at least one eye
* Willing and able to comply with all study related visits and procedures
* In the opinion of the investigator, patients who are appropriate for advanced technology lens implants

Exclusion Criteria:

* History of punctal cautery
* Lacrimal anatomy (e.g., nasolacrimal duct obstruction) that per investigator suggests that the patient would not be a good candidate for lacrimal occlusion or patients for whom lacrimal occlusion would increase risk

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 3- month visit in non-invasive tear break up time (NITBUT) in primary eyes as measured by a non-invasive, automated ocular surface analyzer. | 3 months
  Tear Break-Up time. Tear breakup time (TBUT) is a clinical measurement that assesses the stability of the tear film on the surface of the eye. It measures the time it takes for dry spots to form on the cornea after a complete blink. A rapid breakup indicates tear film instability, which is a common cause of dry eye syndrome.
  Interpreting TBUT results:
  A person's TBUT score is an indicator of their tear film health.
  Normal: A TBUT of 10 seconds or more typically signifies a healthy and stable tear film.
  Marginal/Mild to Moderate Instability: A score of 5 to 9 seconds may suggest mild to moderate tear film instability.
  Low/Dry Eye: A score of less than 5 seconds is a strong indicator of dry eye syndrome caused by tear film dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Kayla Karpuk, OD, Principal Investigator — Vance Thompson Vision Clinic Prof. LLC; Vance Thompson, MD, Principal Investigator — Vance Thompson Vision Clinic Prof. LLC
Locations (1):
- Vance Thompson Vision Clinic, Prof. LLC, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT07155057/Prot_000.pdf
  • Informed Consent Form (2025-08-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT07155057/ICF_001.pdf